CLINICAL TRIAL: NCT02289898
Title: A 3-Arm Phase 2 Double-Blind Randomized Study of Gemcitabine, Abraxane® Plus Placebo Versus Gemcitabine, Abraxane® Plus 1 or 2 Truncated Courses of Demcizumab in Subjects With 1st-Line Metastatic Pancreatic Ductal Adenocarcinoma
Brief Title: Study of Gemcitabine, Abraxane® Plus Placebo Versus Gemcitabine, Abraxane® Plus 1 or 2 Truncated Courses of Demcizumab in Subjects With 1st-Line Metastatic Pancreatic Ductal Adenocarcinoma
Acronym: YOSEMITE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: OncoMed Pharmaceuticals, Inc. (Industry)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Organization: Mereo BioPharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: M18-006
Record Dates: First submitted 2014-11-10; First posted 2014-11-13 (Estimated); Results first posted 2018-08-08 (Actual); Last update posted 2020-09-28 (Actual); Status verified 2020-09

CONDITIONS: Pancreatic Cancer
Keywords: 1st-line metastatic pancreatic ductal adenocarcinoma
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — demcizumab; Albumin-Bound Paclitaxel; Gemcitabine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Abraxane® and gemcitabine plus placebo (Experimental): Abraxane® and gemcitabine plus placebo (3 cycles), Abraxane® and gemcitabine (3 cycles), Abraxane® and gemcitabine plus placebo (3 cycles) and then Abraxane® and gemcitabine until disease progression
  Interventions: Drug: Demcizumab; Drug: Abraxane®; Drug: gemcitabine; Drug: Placebo
- Abraxane® and gemcitabine plus demcizumab plus placebo (Experimental): Abraxane® and gemcitabine plus demcizumab (3 cycles), Abraxane® and gemcitabine (3 cycles), Abraxane® and gemcitabine plus placebo (3 cycles) and then Abraxane® and gemcitabine until disease progression
  Interventions: Drug: Demcizumab; Drug: Abraxane®; Drug: gemcitabine
- Abraxane® and gemcitabine plus demcizumab (Experimental): Abraxane® and gemcitabine plus demcizumab (3 cycles), Abraxane® and gemcitabine (3 cycles), Abraxane® and gemcitabine plus demcizumab (3 cycles) and then Abraxane® and gemcitabine until disease progression
  Interventions: Drug: Demcizumab; Drug: Abraxane®; Drug: gemcitabine

INTERVENTIONS:
Drug: Demcizumab — administered intravenously
Drug: Abraxane® — administered intravenously
Drug: gemcitabine — administered intravenously
Drug: Placebo
  Arms: Abraxane® and gemcitabine plus placebo

SUMMARY:
This is a randomized, double blind, 3 arm (1:1:1) study in subjects with 1st-line metastatic pancreatic ductal adenocarcinoma.

The purpose is to test the efficacy and safety of demcizumab, when given in combination with gemcitabine and Abraxane® compared to placebo. The administration of gemcitabine and Abraxane® is a standard treatment for patients with metastatic pancreatic ductal adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have histologically confirmed metastatic pancreatic ductal adenocarcinoma.. Prior chemotherapy and/or radiotherapy either in the adjuvant or neoadjuvant setting or for metastatic disease is not allowed.
2. Availability of formalin-fixed paraffin-embedded (FFPE) tumor tissue (from either the primary tumor, locoregional disease or a metastatic site), either fresh core-needle-biopsied or archived (two FFPE cores preferred whenever possible). If fresh tissue is obtained, the core biopsy must be done at least 7 days prior to randomization.
3. Age ≥21 years
4. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1 5. Measurable disease per RECIST v1.1
5. Adequate organ and marrow function
6. Signed Informed Consent Form
7. For women of childbearing potential, agreement to use two effective forms of contraception

Exclusion Criteria:

1. Subjects with a neuroendocrine tumor of the pancreas, an acinar tumor of the pancreas or a pancreatic tumor with mixed histologies.
2. Subjects receiving heparin, warfarin, factor Xa inhibitors or other similar anticoagulants. Note: Subjects may be receiving low-dose aspirin and/or non-steroidal anti-inflammatory agents.
3. Subjects with brain metastases, leptomeningeal disease, uncontrolled seizure disorder, or active neurologic disease
4. Subjects with Grade >2 peripheral neuropathy
5. Subjects with clinically significant ascites
6. Malignancies other than pancreatic cancer successfully treated within 3 years prior to randomization, except for adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, treated superficial bladder cancer, localized prostate cancer treated surgically with curative intent, ductal carcinoma in situ treated surgically with curative intent
7. Significant intercurrent illness that will limit the patient's ability to participate in the study or may result in their death over the next 18 months
8. History of a significant allergic reaction attributed to humanized or human monoclonal antibody therapy
9. Subjects with known clinically significant gastrointestinal disease including, but not limited to, inflammatory bowel disease
10. Pregnant women or nursing women
11. Subjects with known HIV infection
12. Known bleeding disorder or coagulopathy

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2015-04-20 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (42):
- United States (22):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Providence Saint Joseph Medical Center, Burbank, California
  - City of Hope, Duarte, California
  - Scripps Cancer Center, La Jolla, California
  - University of California, Davis Comprehensive Cancer Center, Sacramento, California
  - Soulhern California Permanente Medical Group, San Marcos, California
  - Kaiser Permanente Medical Center, Vallejo, California
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Lynn Cancer Institute, Boca Raton, Florida
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kansas Cancer Center, Westwood, Kansas
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - University of Michigan, Ann Arbor, Michigan
  - Dartmouth Hitchcock Medical Center, Norris Cotton Cancer Center, Lebanon, New Hampshire
  - University of Rochester, Rochester, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Kaiser Permanente NW Oncology Research, Portland, Oregon
  - Thomas Jefferson University, Sydney Kimmel Cancer Center, Philadelphia, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - Joe Arrington Cancer Research Treatment Center, Lubbock, Texas
  - Huntsman Cancer Institute at The University of Utah, Salt Lake City, Utah
- Australia (5):
  - Prince of Wales Hospital, Randwick, New South Wales
  - Monash Medical Centre, Moorabbin, Bentleigh East, Victoria
  - Western Health (Sunshine Hospitals), St Albans, Victoria
  - St John of God Murdoch Hospital, Murdoch, Western Australia
  - St. John of God Subiaco Hospital, Subiaco, Western Australia
- Hopital Erasme, Brussels, Brussels Capital, Belgium
- Canada (7):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - British Columbia Cancer Agency, Vancouver, British Columbia
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - London Regional Cancer Program, London, Ontario
  - Sunnybrook Health Sciences Centre, Odette Cancer Centre, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - St Josephs Health Centre, Toronto, Ontario
- Spain (5):
  - Hospital Universitario de Fuenlabrada, Fuenlabrada, Madrid
  - Hospital Universitari Germans Trias i Pujol - lnstituto Catalan d'Oncologia (!CO), Barcelona
  - Hospital General Universitario Gregorio Marafi6n, Madrid
  - Hospital Universitario de Fuenlabrada, Madrid
  - Hospital Universitario Miguel Servet, Zaragoza
- United Kingdom (2):
  - Bristol Haematology & Oncology Centre, Bristol
  - Sarah Cannon Research Institute UK, London

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 207 subjects were randomized and 204 subjects were treated in the study.
Groups:
- Placebo/Placebo Arm: Abraxane and gemcitabine plus placebo (3 cycles), Abraxane and gemcitabine (3 cycles), Abraxane and gemcitabine plus placebo (3 cycles), and then Abraxane and gemcitabine until disease progression.
- Demcizumab/Placebo Arm: Abraxane and gemcitabine plus demcizumab (3 cycles), Abraxane and gemcitabine (3 cycles), Abraxane and gemcitabine plus placebo (3 cycles), and then Abraxane and gemcitabine until disease progression.
- Demcizumab/Demcizumab Arm: Abraxane and gemcitabine plus demcizumab (3 cycles), abraxane and gemcitabine (3 cycles), Abraxane and gemcitabine plus demcizumab (3 cycles), and then Abraxane and gemcitabine until disease progression.
Period: Overall Study
Arm/Group | Placebo/Placebo Arm | Demcizumab/Placebo Arm | Demcizumab/Demcizumab Arm
Started | 68 | 71 | 65
Completed | 16 | 18 | 9
Not Completed | 52 | 53 | 56
Not completed — Death | 5 | 4 | 3
Not completed — Physician Decision | 2 | 5 | 2
Not completed — Withdrawal by Subject | 0 | 4 | 1
Not completed — Adverse Event | 3 | 5 | 5
Not completed — Disease progression | 34 | 28 | 34
Not completed — Use of another anticancer therapy | 0 | 0 | 1
Not completed — Other | 8 | 7 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo/Placebo Arm | Demcizumab/Placebo Arm | Demcizumab/Demcizumab Arm | Total
Number analyzed (Participants) | 68 | 71 | 65 | 204
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 37 | 34 | 30 | 101
  >=65 years | 31 | 37 | 35 | 103
Age, Continuous [Median (Full Range); unit: years] | 62 [41 to 82] | 63 [38 to 85] | 66 [30 to 78] | 63 [30 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 31 | 30 | 88
  Male | 41 | 40 | 35 | 116
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 1 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 1 | 0 | 0 | 1
  White | 60 | 70 | 62 | 192
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 6 | 0 | 1 | 7
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 3 | 5 | 4 | 12
  Belgium | 2 | 2 | 2 | 6
  United States | 17 | 18 | 15 | 50
  United Kingdom | 3 | 2 | 4 | 9
  Australia | 24 | 13 | 19 | 56
  Spain | 19 | 31 | 21 | 71

OUTCOME MEASURES:

1. Primary Outcome: Hazard of Progression in the Placebo/Placebo Arm and the Pooled Demcizumab Arms
Description: Investigator assessed Kaplan-Meier estimates of progression-free survival for placebo/placebo arm and pooled demcizumab arm.
Time Frame: Investigator-assessed progression-free survival time through duration of the study (2 years, 23 days).
Population: Placebo/placebo arm and pooled demcizumab arms (ITT population).
Measure: Count of Participants; unit: Participants
Groups:
- Demcizumab/Placebo and Demcizumab/Demcizumab: Pooled demcizumab arms: Demcizumab/placebo arm - Abraxane and gemcitabine plus demcizumab (3 cycles), Abraxane and gemcitabine (3 cycles), Abraxane and gemcitabine plus placebo (3 cycles), and then Abraxane and gemcitabine until disease progression.
  Demcizumab/demcizumab arn - Abraxane and gemcitabine plus demcizumab (3 cycles), Abraxane and gemcitabine (3 cycles), Abraxane and gemcitabine plus demcizumab (3 cycles), and then Abraxane and gemcitabine until disease progression.
Arm/Group | Placebo/Placebo Arm | Demcizumab/Placebo and Demcizumab/Demcizumab
Number analyzed (Participants) | 68 | 136
Participants
  Progressed (event) | 38 | 70
  Died (event) | 5 | 12
  Censored, follow-up ended | 3 | 7
  Censored, follow-up ongoing | 22 | 47
Statistical Analysis 1: Comparison: Placebo/Placebo Arm vs Demcizumab/Placebo and Demcizumab/Demcizumab; Efficacy (investigator-assessed Kaplan-Meier estimates of progression-free survival) of placebo/placebo arm to the pooled demcizumab arm (i.e., placebo/placebo arm to demcizumab/placebo and demcizumab/demcizumab arms) in subjects with first-line metastatic pancreatic ductal adenocarcinoma; Test type: Superiority; p = 0.7158, Wilcoxon (Mann-Whitney); Hazard Ratio (HR) = .930, 95% CI 2-sided [0.630 to 1.375]

ADVERSE EVENTS:
Time Frame: Adverse event data are collected from the time of randomization through 30 days after discontinuation from the study (30 dates from the date of the treatment termination visit). Total study duration: 2 years, 23 days.
Arm/Group | Placebo/Placebo Arm | Demcizumab/Placebo Arm | Demcizumab/Demcizumab Arm
All-Cause Mortality (participants affected / at risk) | 5/68 | 12/71 | 3/65
Serious Adverse Events (participants affected / at risk) | 40/68 | 49/71 | 34/65
Other Adverse Events (participants affected / at risk) | 68/68 | 71/71 | 65/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo/Placebo Arm (N=68) | Demcizumab/Placebo Arm (N=71) | Demcizumab/Demcizumab Arm (N=65)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Tumour rupture (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 6 (6) | 3 (3) | 6 (6)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 1 (1) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Anaesthetic complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Liver function test increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (4) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 2 (2)
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0)
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Generalised tonic-clonic seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Peroneal nerve palsy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 1 (1)
Papilloedema (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 5 (5) | 4 (4) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 4 (4) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 0 (0) | 3 (3)
Nausea (Gastrointestinal disorders) | 4 (4) | 1 (1) | 2 (2)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2)
Ascites (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Colonic fistula (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diverticular perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intestinal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatic duct obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pancreatic insufficiency (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 1 (1) | 1 (1) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0)
Bile duct obstruction (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatic haematoma (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Jaundice (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 3 (3)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Device dislocation (Product Issues) | 0 (0) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Vertebral lesion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 3 (3) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Food intolerance (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 3 (3) | 4 (4) | 4 (4)
Liver abscess (Infections and infestations) | 2 (2) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Abdominal abscess (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Bacterial infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bacterial sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Colonic abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Hepatic infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Tick-borne fever (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo/Placebo Arm (N=68) | Demcizumab/Placebo Arm (N=71) | Demcizumab/Demcizumab Arm (N=65)
Hypertension (Vascular disorders) | 10 (10) | 17 (17) | 21 (21)
Hypotension (Vascular disorders) | 11 (11) | 6 (6) | 5 (5)
Deep vein thrombosis (Vascular disorders) | 7 (7) | 4 (4) | 9 (9)
Fatigue (General disorders) | 34 (34) | 31 (31) | 37 (37)
Oedema peripheral (General disorders) | 29 (29) | 39 (39) | 34 (34)
Pyrexia (General disorders) | 24 (24) | 30 (30) | 23 (23)
Asthenia (General disorders) | 18 (18) | 27 (27) | 20 (20)
Chills (General disorders) | 6 (6) | 3 (3) | 8 (8)
Headache (General disorders) | 12 (12) | 13 (13) | 22 (22)
Insomnia (Psychiatric disorders) | 9 (9) | 8 (8) | 9 (9)
Anxiety (Psychiatric disorders) | 10 (10) | 5 (5) | 3 (3)
Depression (Psychiatric disorders) | 6 (6) | 3 (3) | 7 (7)
Platelet count decreased (Investigations) | 16 (16) | 20 (20) | 13 (13)
Alanine aminotransferase increased (Investigations) | 16 (16) | 15 (15) | 15 (15)
Neutrophil count decreased (Investigations) | 16 (16) | 12 (12) | 12 (12)
Aspartate aminotransferase increased (Investigations) | 13 (13) | 5 (5) | 12 (12)
Brain natriuretic peptide increased (Investigations) | 5 (5) | 11 (11) | 14 (14)
White blood cell count decreased (Investigations) | 9 (9) | 4 (4) | 10 (10)
Blood alkaline phosphatase increased (Investigations) | 5 (5) | 6 (6) | 10 (10)
Weight decreased (Investigations) | 8 (8) | 5 (5) | 8 (8)
Blood bilirubin increased (Investigations) | 6 (6) | 3 (3) | 3 (3)
Gamma-glutamyltransferase increased (Investigations) | 5 (5) | 2 (2) | 5 (5)
Anaemia (Blood and lymphatic system disorders) | 27 (27) | 43 (43) | 35 (35)
Thrombocytopenia (Blood and lymphatic system disorders) | 15 (15) | 14 (14) | 16 (16)
Neutropenia (Blood and lymphatic system disorders) | 21 (21) | 24 (24) | 25 (25)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 18 (18) | 16 (16) | 10 (10)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 13 (13) | 17 (17)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 12 (12) | 11 (11)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4) | 8 (8)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 7 (7) | 7 (7)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2) | 5 (5)
Dysgeusia (Nervous system disorders) | 18 (18) | 16 (16) | 17 (17)
Peripheral sensory neuropathy (Nervous system disorders) | 16 (16) | 17 (17) | 17 (17)
Dizziness (Nervous system disorders) | 10 (10) | 5 (5) | 7 (7)
Neurotoxicity (Nervous system disorders) | 2 (2) | 11 (11) | 4 (4)
Vision blurred (Eye disorders) | 3 (3) | 3 (3) | 5 (5)
Nausea (Gastrointestinal disorders) | 42 (42) | 38 (38) | 41 (41)
Diarrhoea (Gastrointestinal disorders) | 34 (34) | 41 (41) | 45 (45)
Vomiting (Gastrointestinal disorders) | 27 (27) | 32 (32) | 25 (25)
Constipation (Gastrointestinal disorders) | 20 (20) | 21 (21) | 28 (28)
Abdominal pain (Gastrointestinal disorders) | 24 (24) | 16 (16) | 27 (27)
Stomatitis (Gastrointestinal disorders) | 13 (13) | 12 (12) | 15 (15)
Abdominal pain upper (Gastrointestinal disorders) | 13 (13) | 6 (6) | 8 (8)
Dry mouth (Gastrointestinal disorders) | 7 (7) | 9 (9) | 6 (6)
Ascites (Gastrointestinal disorders) | 9 (9) | 6 (6) | 3 (3)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 6 (6) | 7 (7) | 5 (5)
Abdominal distension (Gastrointestinal disorders) | 5 (5) | 4 (4) | 4 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 30 (30) | 33 (33) | 28 (28)
Rash (Skin and subcutaneous tissue disorders) | 18 (18) | 14 (14) | 17 (17)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (4) | 5 (5) | 5 (5)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 (6) | 3 (3) | 5 (5)
Erythema (Gastrointestinal disorders) | 3 (3) | 7 (7) | 3 (3)
Hypokalaemia (Gastrointestinal disorders) | 7 (7) | 7 (7) | 6 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 16 (16) | 10 (10) | 13 (13)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (6) | 10 (10) | 15 (15)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (8) | 9 (9) | 10 (10)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 (8) | 5 (5) | 7 (7)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3) | 6 (6)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (2) | 4 (4)
Decreased appetite (Metabolism and nutrition disorders) | 19 (19) | 30 (30) | 27 (27)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 8 (8) | 10 (10) | 9 (9)
Dehydration (Metabolism and nutrition disorders) | 6 (6) | 10 (10) | 6 (6)
Hyperglycaemia (Metabolism and nutrition disorders) | 11 (11) | 5 (5) | 4 (4)
Hyponatraemia (Metabolism and nutrition disorders) | 6 (6) | 4 (4) | 8 (8)
Hypophosphataemia (Metabolism and nutrition disorders) | 5 (5) | 5 (5) | 6 (6)
Hypocalcaemia (Metabolism and nutrition disorders) | 6 (6) | 7 (7) | 2 (2)
Urinary tract infection (Infections and infestations) | 7 (7) | 5 (5) | 7 (7)
Upper respiratory tract infection (Infections and infestations) | 6 (6) | 6 (6) | 6 (6)
Oral candidiasis (Infections and infestations) | 8 (8) | 2 (2) | 4 (4)
Cellulitis (Infections and infestations) | 6 (6) | 5 (5) | 1 (1)
Sepsis (Infections and infestations) | 3 (3) | 5 (5) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-03-08): https://cdn.clinicaltrials.gov/large-docs/98/NCT02289898/SAP_000.pdf
  • Study Protocol and Informed Consent Form (2016-12-19): https://cdn.clinicaltrials.gov/large-docs/98/NCT02289898/Prot_ICF_001.pdf